CLINICAL TRIAL: NCT03944187
Title: Sonographic Assessment of Fetal Head Circumference, Cervical Length and Fetal Head to Cervix Angle for Prediction of Labor Induction Success
Brief Title: Sonographic Assessment for Prediction of Labor Induction Success
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0529-18-RMB
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal sonography — Transvaginal sonography for measurement of cervical length, fetal head circumference and fetal head to cervix angle .

SUMMARY:
The study is conducted to assess several sonographic parameters for prediction of labor induction success. These parameters include cervical length, fetal head circumference, and fetal head to cervix angle.

DETAILED DESCRIPTION:
Pregnant women at term over 37 weeks' gestation visiting the obstetric emergency room for various obstetric indications will be assessed. Women with obstetric or medical indication for induction will receive an explanation regarding the study protocol and will sign an informed consent.

After recruitment and during the evaluation in the obstetric emergency room, patients will undergo transvaginal sonography during which, cervical length, fetal head circumference and fetal head to cervix angle will be measured.

Relevant demographic and obstetric information will be collected from a computerized database.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Term pregnancy.

Exclusion Criteria:

* Multiple gestation.
* Fetal anomalies and malformations.
* Preterm pregnancy.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women with singleton pregnancy over 37 weeks' gestation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Success in induction of labor | From admission to the obstetric emergency room up to 24 hours postpartum
  Vaginal delivery rate after labor induction

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No